CLINICAL TRIAL: NCT03944655
Title: Does Strepsils® With Lignocaine Lozenges Reduce Post Operative Sore Throat Due To Supraglottic Airway Devices
Acronym: POSTrepsils
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr Sebastian Sundaraj (Other)
Responsible Party: Sponsor-Investigator, Dr Sebastian Sundaraj, Sponsor-Investigator, University of Malaya
Organization: University of Malaya (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 201887-6582
Record Dates: First submitted 2019-05-05; First posted 2019-05-09 (Actual); Last update posted 2020-01-28 (Actual); Status verified 2020-01

CONDITIONS: Sore Throat; Post Operative Sore Throat
Keywords: Post operative sore throat; Post operative dysphagia; Post operative dysphonia
MeSH Terms: conditions — Pharyngitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Strepsils (Active Comparator)
  Interventions: Drug: Strepsils Anaesthetic Formula
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Clear Mint Drops

INTERVENTIONS:
Drug: Strepsils Anaesthetic Formula — Oral administration of a Strepsils® Max Plus lozenge containing the active ingredients amylmetacresol 0.6 mg, 2,4-dichlorobenzyl alcohol 1.2 mg, lignocaine hydrochloride 10mg with sweeteners and flavourings.
  Other Names: Strepsils Max Plus
  Arms: Strepsils
Dietary Supplement: Clear Mint Drops — Oral administration of a lozenge containing glucose syrup, sugar, and flavourings
  Arms: Placebo

SUMMARY:
The primary objective of this study is to assess the effect of preoperative administration of oral Strepsils® with added Lignocaine lozenges on the incidence of postoperative sore throat (POST) after general anaesthesia using a Supraglottic Airway Device (SAD).

Patients undergoing surgery with general anaesthesia will require ventilation of their lungs with either a flexible tube placed beyond the voice box called an endotracheal tube (ETT) or a tube placed above the voice box called a Supraglottic Airway Device. This tube helps oxygenate the patient and delivers anaesthetic gas to the lungs.

The procedure is invasive and uncomfortable, and one of the most common complaints is a sore and inflamed throat after the tube is taken out. This is termed postoperative sore throat (POST). The incidence of POST after SAD is comparable with the ETT and though many studies have focused on ETT, few have examined the SAD.

After written informed consent is received in pre-op, a sealed and coded envelope with either the Strepsils lozenges or the placebo lozenges will be given to the patient to be administered orally, with the instruction to dissolve the lozenge by sucking on it 45 minutes prior to surgery. Upon completion of surgery and emergence from general anaesthesia, the patient will be assessed regarding the incidence and severity of sore throat, difficulty in swallowing and difficulty in speaking by the investigator using an interview format. The severity of these symptoms will be graded on a 4-point scale ranging from 0 to 3; 0 being no symptoms, 1 being mild symptoms, 2 being moderate symptoms, and 3 being severe symptoms. This evaluation will be performed at 30 minutes and 24 hours post removal of SAD.

DETAILED DESCRIPTION:
The incidence of postoperative sore throat (POST) has been reported up to 62% following general anaesthesia with varying severity from mild to severe. It is among the top undesirable events experienced by patients after anaesthesia. The supraglottic airway device (SAD) is commonly used as an airway device during the delivery of general anaesthesia. The incidence of POST after SAD use has been documented of up to 49% and is comparable with the incidence of up to 45% when using an endotracheal tube (ETT).

Many studies have been evaluating the occurrence of POST with the use of an ETT but studies investigating POST and the use of SAD are limited. A recent study comparing sore throat following three SADs (LMA™ Unique, LMA™ Supreme and I-gel®) found that the incidence of POST was not significantly different between any of them.

There are various drugs being extensively investigated to reduce the incidence and severity of POST such as Lignocaine, Dexamethasone, NSAIDs, Liquorice and NMDA receptor antagonists [1]. A Cochrane review on the use of Lignocaine for endotracheal intubation concluded that Lignocaine applied topically or administered systemically resulted in reduced risk and severity of POST.

Amylmetacresol and Dichlorobenzyl Alcohol, the active ingredient in the standard preparation of Strepsils® lozenges has been shown to reduce the intensity of sore throat in non-anaesthetised subjects, including one study involving Strepsils® Max Plus lozenges which additionally contains Lignocaine, a local anaesthetic agent. Currently studies that evaluated POST after endotracheal intubation using the standard preparation of Strepsils® (without Lignocaine) have reported a reduction in the incidence and severity of POST.

The effect of Strepsils® Max Plus (with Lignocaine) lozenges on POST and particularly due to SAD is not known and is the basis of this study. It is the investigator's hypothesis that Strepsils® with added Lignocaine will reduce the incidence and severity of POST based on existing studies that showed the individual and combined beneficial effect of both substances.

The goal of this study is to identify a simple, safe, and inexpensive perioperative intervention to reduce the incidence and severity of post operative sore throat due to supraglottic airway devices.

Eligible participants include adult patients scheduled to undergo elective surgery under general anaesthesia using a supraglottic airway device. This study is a prospective, randomised, double-blinded study involving 60 subjects and they will assessed on the incidence and severity of sore throat, dysphagia and dysphonia at 30 minutes and 24 hours after removal of the supraglottic airway device using an interview format.

Outcomes from this study can be extended to patients who will be receiving general anaesthesia using a supraglottic airway device in the future.

ELIGIBILITY:
Inclusion Criteria:

* Greater than 18 years of age
* American Society of Anesthesiologists Class I-II
* Supraglottic Airway Device usage duration < 2 hours

Exclusion Criteria:

* History of upper respiratory tract infection, sore throat, dysphonia, or dysphagia in the past 2 weeks
* Morbidly obese (body mass index >35 kg/m2)
* Increased risk of regurgitation or aspiration (eg. symptomatic gastro-oesophageal reflux, hiatus hernia)
* Pregnant or nursing
* Known allergies to study drug
* More than one attempt at Supraglottic Airway Device insertion or use of adjuncts during insertion
* Insertion/presence of a gastric tube
* Expected airway difficulties or conversion to endotracheal tube

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2019-01-17 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
Incidence of sore throat | 30 minutes after the removal of Supraglottic Airway Device
  Presence of sore throat defined as constant pain, independent of swallowing
Incidence of sore throat | 24 hours after the removal of Supraglottic Airway Device
  Presence of sore throat defined as constant pain, independent of swallowing

SECONDARY OUTCOMES:
Severity of sorethroat | 30 minutes after the removal of Supraglottic Airway Device
  Severity will be graded by the patient as 0=null; 1=mild; 2=moderate; 3=severe
Severity of sorethroat | 24 hours after the removal of Supraglottic Airway Device
  Severity will be graded by the patient as 0=null; 1=mild; 2=moderate; 3=severe
Incidence of dysphagia | 30 minutes after the removal of Supraglottic Airway Device
  Presence of dysphagia defined as difficulty or pain provoked by swallowing
Incidence of dysphagia | 24 hours after the removal of Supraglottic Airway Device
  Presence of dysphagia defined as difficulty or pain provoked by swallowing
Incidence of dysphonia | 30 minutes after the removal of Supraglottic Airway Device
  Presence of dysphonia defined as difficulty or pain on speaking
Incidence of dysphonia | 24 hours after the removal of Supraglottic Airway Device
  Presence of dysphonia defined as difficulty or pain on speaking
Severity of dysphagia | 30 minutes after the removal of Supraglottic Airway Device
  Severity will be graded by the patient as 0=null; 1=mild; 2=moderate; 3=severe
Severity of dysphagia | 24 hours after the removal of Supraglottic Airway Device
  Severity will be graded by the patient as 0=null; 1=mild; 2=moderate; 3=severe
Severity of dysphonia | 30 minutes after the removal of Supraglottic Airway Device
  Severity will be graded by the patient as 0=null; 1=mild; 2=moderate; 3=severe
Severity of dysphonia | 24 hours after the removal of Supraglottic Airway Device
  Severity will be graded by the patient as 0=null; 1=mild; 2=moderate; 3=severe
Adverse effects of study drug | 30 minutes after the removal of Supraglottic Airway Device
  Any untoward medical occurrence in a subject administered an investigational product and which does not necessarily have a causal relationship with treatment.
Adverse effects of study drug | 24 hours after the removal of Supraglottic Airway Device
  Any untoward medical occurrence in a subject administered an investigational product and which does not necessarily have a causal relationship with treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian Sundaraj, MD, Principal Investigator — University of Malaya
Locations (1):
- University Malaya Medical Centre, Kuala Lumpur, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] El-Boghdadly K, Bailey CR, Wiles MD. Postoperative sore throat: a systematic review. Anaesthesia. 2016 Jun;71(6):706-17. doi: 10.1111/anae.13438. Epub 2016 Mar 28. PMID 27158989
- [Background] Macario A, Weinger M, Carney S, Kim A. Which clinical anesthesia outcomes are important to avoid? The perspective of patients. Anesth Analg. 1999 Sep;89(3):652-8. doi: 10.1097/00000539-199909000-00022. PMID 10475299
- [Background] Higgins PP, Chung F, Mezei G. Postoperative sore throat after ambulatory surgery. Br J Anaesth. 2002 Apr;88(4):582-4. doi: 10.1093/bja/88.4.582. PMID 12066737
- [Background] Wong DT, Tam AD, Mehta V, Raveendran R, Riad W, Chung FF. New supraglottic airway with built-in pressure indicator decreases postoperative pharyngolaryngeal symptoms: a randomized controlled trial. Can J Anaesth. 2013 Dec;60(12):1197-203. doi: 10.1007/s12630-013-0044-2. Epub 2013 Oct 5. PMID 24097301
- [Background] L'Hermite J, Dubout E, Bouvet S, Bracoud LH, Cuvillon P, Coussaye JE, Ripart J. Sore throat following three adult supraglottic airway devices: A randomised controlled trial. Eur J Anaesthesiol. 2017 Jul;34(7):417-424. doi: 10.1097/EJA.0000000000000539. PMID 27755181
- [Background] Tanaka Y, Nakayama T, Nishimori M, Tsujimura Y, Kawaguchi M, Sato Y. Lidocaine for preventing postoperative sore throat. Cochrane Database Syst Rev. 2015 Jul 14;2015(7):CD004081. doi: 10.1002/14651858.CD004081.pub3. PMID 26171894
- [Background] Weckmann G, Hauptmann-Voss A, Baumeister SE, Klotzer C, Chenot JF. Efficacy of AMC/DCBA lozenges for sore throat: A systematic review and meta-analysis. Int J Clin Pract. 2017 Oct;71(10). doi: 10.1111/ijcp.13002. Epub 2017 Sep 4. PMID 28869700
- [Background] Ebneshahidi A, Mohseni M. Strepsils(R) tablets reduce sore throat and hoarseness after tracheal intubation. Anesth Analg. 2010 Oct;111(4):892-4. doi: 10.1213/ANE.0b013e3181d00c60. Epub 2010 Feb 8. PMID 20142339
- [Background] Gupta D, Agrawal S, Sharma JP. Evaluation of preoperative Strepsils lozenges on incidence of postextubation cough and sore throat in smokers undergoing anesthesia with endotracheal intubation. Saudi J Anaesth. 2014 Apr;8(2):244-8. doi: 10.4103/1658-354X.130737. PMID 24843341
- [Background] Smith I, Kranke P, Murat I, Smith A, O'Sullivan G, Soreide E, Spies C, in't Veld B; European Society of Anaesthesiology. Perioperative fasting in adults and children: guidelines from the European Society of Anaesthesiology. Eur J Anaesthesiol. 2011 Aug;28(8):556-69. doi: 10.1097/EJA.0b013e3283495ba1. PMID 21712716
- [Background] Ouanes JP, Bicket MC, Togioka B, Tomas VG, Wu CL, Murphy JD. The role of perioperative chewing gum on gastric fluid volume and gastric pH: a meta-analysis. J Clin Anesth. 2015 Mar;27(2):146-52. doi: 10.1016/j.jclinane.2014.07.005. Epub 2014 Nov 28. PMID 25442242
- [Background] Bouvet L, Loubradou E, Desgranges FP, Chassard D. Effect of gum chewing on gastric volume and emptying: a prospective randomized crossover study. Br J Anaesth. 2017 Nov 1;119(5):928-933. doi: 10.1093/bja/aex270. PMID 29077816
- [Background] Timmermann A, Bergner UA, Russo SG. Laryngeal mask airway indications: new frontiers for second-generation supraglottic airways. Curr Opin Anaesthesiol. 2015 Dec;28(6):717-26. doi: 10.1097/ACO.0000000000000262. PMID 26539790